CLINICAL TRIAL: NCT03553433
Title: A Phase 4 Multicenter, Randomized, Placebo-controlled Study Evaluating the Effect of Apremilast on Pruritus and Quality of Life of Patients With Moderate-to-severe Scalp Psoriasis
Brief Title: Apremilast Treatment for Pruritus and Quality of Life in Scalp Psoriasis
Acronym: APRESCALP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DER-USZ-AAN-021
Record Dates: First submitted 2018-04-18; First posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Psoriasis of Scalp; Psoriasis Vulgaris
Keywords: apremilast; quality of life; pruritus; oral drug; placebo
MeSH Terms: conditions — Pruritus | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Experimental): Apremilast 30mg bd
  Interventions: Drug: Apremilast 30mg
- Placebo Oral Tablet (Placebo Comparator): Excipiens
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Apremilast 30mg — Anti-psoriatic drug
  Other Names: Otezla
  Arms: Verum
Drug: Placebo Oral Tablet — Indistinguishable tablets not containing apremilast, Placebo Oral Tablet
  Other Names: Placebo
  Arms: Placebo Oral Tablet

SUMMARY:
A phase 4 multicenter, randomized, placebo-controlled Study evaluating the Effect of Apremilast on Pruritus and Quality of Life of Patients with moderate-to-severe Scalp Psoriasis

DETAILED DESCRIPTION:
The scalp is the most frequently affected body region in psoriasis. Scalp Psoriasis can impair the quality of life greatly due to pruritus. This is however not usually investigated as a primary outcome of treatments.

This study will investigate the effects of apremilast on the pruritus and quality of life and other patient reported outcomes in patients with scalp psoriasis.

ELIGIBILITY:
Inclusion criteria:

1. Adult (>18yrs);
2. Signed informed consent
3. Clinical diagnosis of chronic plaque psoriasis for at least 3 months as determined by the subject's medical history and confirmation of diagnosis through physical examination by the Investigator;
4. Psoriatic lesions with DLQI >10 and involvement of >20% of the scalp and pruritus with a VAS score of > 50 (0-100);
5. Candidate for systemic therapy;
6. Females who are of child-bearing potential should be practicing birth control throughout the study and for 70 days after the last dose of study drug;
7. Subject is judged to be in good health as determined by the Investigator based upon the results of medical history, laboratory profile and physical examination.
8. Creatinine < 80 umol/l at Inclusion

Exclusion criteria:

1. Erythrodermic Ps, medication-induced or medication-exacerbated Ps or new onset guttate Ps or other skin conditions at the time of the screening visit (e.g. eczema) that would interfere with evaluations of the effect of the investigational product on Ps;
2. Use of any anti-psoriatic therapy last administered less than 4 weeks of start of study drug such as

   1. Three months or 5 PK half-lives, whichever is longer, for biologics tumor necrosis factor (TNF) antagonists, interleukin (IL) 12/23/17 inhibitors or other biologic drugs
   2. 4 weeks for immunosuppressive / -modulating drugs including cyclosporine A, methotrexate, azathioprine, mycophenolate mofetil, fumaric acid esters, retinoids, JAK inhibitors, corticosteroids, any other experimental drug, etc.
   3. Topical medications (eg. Corticosteroids) except coal tar shampoo, and/or salicylic acid scalp preparations on scalp lesions.
   4. 4 weeks for phototherapy (ie, UVB, PUVA).
3. Infection(s) requiring treatment with intravenous (IV) anti-infectives within 30 days prior to the Baseline visit or oral anti-infectives within 14 days prior to the Baseline visit;
4. Positive serology for hepatitis B, hepatitis C, HIV indicating acute or chronic infection;
5. Chronic recurring bacterial infections or active TB;
6. Positive pregnancy test at Screening or at the Baseline visit;
7. Female subjects who are pregnant or breast-feeding or considering becoming pregnant during the study;
8. History of clinically significant alcohol or drug abuse in the last 12 months;
9. Known hypersensitivity to the excipients of Otezla® as stated in the label;
10. Subject is considered by the Investigator, for any reason, to be an unsuitable candidate for the study.
11. Prior history of suicide attempt at any time in the subject's life time prior to signing the informed consent and randomization, or major psychiatric illness requiring hospitalization within the last 3 years prior to signing the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Scalp VAS Pruritus assessment | Weeks 16
  Pruritus VAS Scale (0 - 100)

SECONDARY OUTCOMES:
Scalp VAS Pruritus assessment | Weeks 0, 4, 32, 52
  Pruritus VAS Scale (0 - 100)
% BSA | Weeks 0, 4, 16, 32, 52
  Body surface area
% BSA of scalp | Weeks 0, 4, 16, 32, 52
  Body surface area of scalp
PrecisePASI | Weeks 0, 4, 16, 32, 52
  Psoriasis Area and Severity Index, modified to measure in percentages
PGA | Weeks 0, 4, 16, 32, 52
  Physicians Global Assessment (0 - 5)
Scalp-PGA | Weeks 0, 4, 16, 32, 52
  Physicians Global Assessment of the Scalp (0 - 5)
DLQI | Weeks 0, 4, 16, 32, 52
  Skin related Quality of life (0 to 30)
Scalpdex | Weeks 0, 4, 16, 32, 52
  23 items related to scalp symptoms
PSSI | Weeks 0, 4, 16, 32, 52
  Psoriasis score measuring intensity on the scalp
VAS pruritus assessment | Weeks 0, 4, 16, 32, 52
  Pruritus VAS Scale (0 - 100)
EQ-5D | Weeks 0, 4, 16, 32, 52
  Health-related Quality of Life Instrument

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Navarini, MD PhD, Principal Investigator — University of Zurich
Locations (4):
- Switzerland (4):
  - KSSG, Sankt Gallen, Canton of St. Gallen
  - Inselspital, Bern
  - CHUV, Lausanne
  - Department of Dermatology, University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No